CLINICAL TRIAL: NCT06611436
Title: BeCoMe-9: A Phase 1/2 Dose Escalation and Expansion Study of BE-101 for the Treatment of Adults With Moderately Severe or Severe Hemophilia B
Brief Title: BeCoMe-9: A Clinical Study of BE-101 for the Treatment of Adults With Moderately Severe or Severe Hemophilia B
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Be Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BE-101-01
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia B; Hemophilia B, Moderately Severe or Severe
Keywords: Hemophilia B; Dose Escalation
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 - Dose Escalation, Dose Level 1 (Experimental)
  Interventions: Drug: BE-101
- Part 1 - Dose Escalation, Dose Level 2 (Experimental)
  Interventions: Drug: BE-101
- Part 1 - Dose Escalation, Dose Level 3 (Experimental)
  Interventions: Drug: BE-101
- Part 2 - Dose Expansion, Cohort 2a Adult Expansion, Optimal Dose Selected in Part 1 Dose Escalation (Experimental)
  Interventions: Drug: BE-101

INTERVENTIONS:
Drug: BE-101 — IV Infusion of BE-101 dose from Dose Level 1
  Arms: Part 1 - Dose Escalation, Dose Level 1
Drug: BE-101 — IV Infusion of BE-101 dose from Dose Level 2
  Arms: Part 1 - Dose Escalation, Dose Level 2
Drug: BE-101 — IV Infusion of BE-101 dose from Dose Level 3
  Arms: Part 1 - Dose Escalation, Dose Level 3
Drug: BE-101 — IV Infusion of BE-101 with optimal dose selected from Part 1 Dose Escalation
  Arms: Part 2 - Dose Expansion, Cohort 2a Adult Expansion, Optimal Dose Selected in Part 1 Dose Escalation

SUMMARY:
The BeCoMe-9 Study (BE-101-01) is a Phase 1/2, first in human, multi-center, open-label, dose-escalation study to evaluate the safety and clinical activity of a single intravenous (IV) dose of BE-101 in adults with moderately severe or severe Hemophilia B. Once infused, BE-101 is designed to engraft and continuously secrete FIX into the circulation to restore clinically meaningful levels of active FIX. BE-101 is an autologous (person's own cells) B Cell Medicine (BCM) which uses CRISPR/Cas9 gene editing to precisely insert human FIX gene into those cells.

DETAILED DESCRIPTION:
The study includes 2 distinct parts: Part 1 and Part 2. In Part 1, an ascending-dose design will be utilized to enable evaluation of increasing doses in a stepwise manner. The objective for this dose escalation is to identify the dose of BE-101 required to achieve desired FIX activity 28 days after infusion. Upon identification of a safe and efficacious dose in Part 1, an expansion phase (Part 2) will initiate. The initial cohort in the Part 2 expansion (Part 2a) phase will include up to 6 adult participants to further characterize the safety and activity of BE-101 at the selected dose. Additional cohorts for adolescents and redosing for participants in Part 1 of the study will occur following data availability of Part 1.

Up to 24 participants will be enrolled across Part 1 (up to 18) and Part 2a (up to 6). Consented participants will complete a screening period to assess eligibility and upon enrollment will undergo leukapheresis collection to support BE-101 manufacturing. Following administration, participants will be monitored for safety and clinical activity. The total duration of study participation is approximately 52 weeks post IV administration of BE-101.

ELIGIBILITY:
Inclusion Criteria:

* Adult Males (≥18) with moderately severe to severe Hemophilia B (FIX deficiency)
* Received ≥50 exposure days to Factor IX products preceding enrollment.
* Currently receiving prophylaxis treatment
* Adequate organ function and clinical labs
* Able to tolerate study procedures including leukapheresis.

Exclusion Criteria:

* Pre-existing or history of specific diseases

  * B-Cell malignancy, EBV lymphoproliferative disease
  * Primary immunodeficiency disease or disorder (PIDD) or systemic immuno-suppression
  * Arterial and/or venous thromboembolic events within 2 years prior to dosing
  * History of anaphylaxis or nephrotic syndrome
  * Active infection (HIV, Hep B or C)
* History of inhibitor to FIX or inhibitor
* History of an allergic reaction or anaphylaxis to FIX products
* Planned surgical procedure within 6 months from BE-101 administration
* Previously dosed with gene therapy
* Participated in an interventional study and/or received an interventional study drug within 30 days or five-half-lives (whichever is longer) of consent into BeCoMe-9 and for the duration of the study
* Planned participation in clinical trial within one year after BE-101
* Administration of an investigational agent or vaccine within 28 days of leukapheresis and dosing of BE-101

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) and Serious Adverse Events (SAEs) | 1 year post dose
  Incidence of AEs and SAEs

SECONDARY OUTCOMES:
FIX Activity | Baseline to 1 year post dose
  Change From Baseline in FIX Activity
Annualized Bleed Rate (ABR) | 1 year post dose
  ABR (spontaneous and traumatic) for all bleeds. Annualized bleed rates overall and by severity will be presented.
Bleeding Episodes | 1 year post dose
  Number of bleeding episodes (total, spontaneous, and traumatic). Bleeding episodes will be summarized by subject and overall, and will include number, duration, and severity.
Target Joints | 1 year post dose
  Number of target joints. A target joint is defined as a major joint (e.g. hip, elbow, wrist, shoulder, knee, ankle) into which repeated bleeding occurs (frequency of 3 or more bleeding episodes into the same joint in a consecutive 12 week period) and with symptoms of pre-existing target joint involvement (eg, synovitis, persistent swelling, effusion, limitation of range of motion).
FIX Antigen Concentration | Baseline to 1 year post dose
  Change From Baseline in FIX Antigen concentration
Exogenous FIX Concentrate | 1 year post dose
  Number of infusions of exogenous FIX concentrate
FIX Replacement Therapy | 1 year post dose
  Total consumption of exogenous FIX replacement therapy (IU) after BE-101 administration
FIX Inhibitor | 1 year post dose
  FIX inhibitor development post BE-101 administration

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California, Davis, Davis, California
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington Center for Bleeding Disorders, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No